CLINICAL TRIAL: NCT00216619
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Trial to Investigate the Efficacy and Tolerability of Topiramate in Prolonged Migraine Prevention
Brief Title: The Prolonged Use of Topiramate for Preventing Migraine Headaches
Acronym: PROMPT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003931; 2005-000321-29 (EudraCT Number); TOPMAT-MIG-303 (Other: Janssen CTMS ID)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Migraine
Keywords: chronic migraine; Topiramate; migraine; headache; chronic headache
MeSH Terms: conditions — Migraine Disorders; Headache; Headache Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Label Phase (Experimental): Topiramate treatment started with one tablet per day, taken in the evening, for the first 7 days of the OL phase. Each tablet contained 25 mg topiramate. After one week, the dose was raised to two tablets per day: one tablet was taken in the morning, the other in the evening. Until Week 26
  Interventions: Drug: Topiramate
- Double Blind and Roll Out Phase (Experimental): the trial medication consisted of topiramate 25 mg tablets or matching placebo tablets which were identical in appearance, taste and smell. DB randomisation phase (after the 26-weeks OL phase) were randomly allocated (1:1) to one of the two treatment groups (topiramate or placebo). The randomisation took place at Visit 6 (Week 26).
  Interventions: Drug: Topiramate; Drug: Topiramate - Placebo

INTERVENTIONS:
Drug: Topiramate — topiramate treatment started with one tablet per day, taken in the evening, for the first 7 days of the OL phase. Each tablet contained 25 mg topiramate. After one week, the dose was raised to two tablets per day: one tablet was taken in the morning, the other in the evening.
Drug: Topiramate - Placebo — the trial medication consisted of topiramate 25 mg tablets or matching placebo tablets which were identical in appearance, taste and smell. DB randomisation phase (after the 26-weeks OL phase) were randomly allocated (1:1) to one of the two treatment groups (topiramate or placebo). The randomisation took place at Visit 6 (Week 26)
  Arms: Double Blind and Roll Out Phase

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness (beyond 6 months) of individualized doses (100 to 200 milligrams) of topiramate for the prevention of migraine headaches over a period of 26 weeks.

DETAILED DESCRIPTION:
Previous studies have shown that topiramate is effective in preventing migraine headaches. This study will start with a 4-week baseline period in which no treatment is given, followed by a 26-week period in which each patient's dose is adjusted and then kept stable for 4 weeks. The dose will start at 25 milligrams of topiramate per day and will be increased 25 milligrams per day once weekly and then raised to either the target--100 milligrams per day--or the maximum dose that is well tolerated up to 200 milligrams per day. Patients randomized to receive topiramate will remain on that dose. The comparison phase of the study is a 26-week period in which the change in migraine days of patients on topiramate (taking at least 50 milligrams per day) is compared with the change in migraine days for patients on the placebo. Also studied will be the patients' health-related quality of life as assessed by questionnaires filled out at specific visits as well as the patients' views of the safety and tolerability of topiramate. The study hypothesis is that the number of migraine days, periods, and attacks during the last 4 weeks of the double-blind phase, relative to the last 4 weeks of the open-label phase, is reduced more in the topiramate group than the placebo group. During open-label (26-weeks) and double-blind phase (26-weeks), patients receiving topiramate will take 25 milligrams to 100 milligrams daily by mouth; increased by 25 milligrams per day once weekly; dose cannot exceed 200 milligrams per day and must be stable for the last 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Established history of migraine for at least one year;
* Migraine meets HIS (International Headache Society) criteria
* An average of at least 4 monthly migraine days during the 3 months preceding trial entry
* Capable of keeping trial records; Exclusion Criteria:
* Patient used migraine prophylactic medication in the month prior to trial entry (flunarizine: 3 months prior to entry)
* Patient had failed (lack of efficacy) more than two adequate previous regimens of migraine prophylactic medications
* Patient had a history of severe drug allergy or hypersensitivity
* Patient overused analgesics, opiates, ergots and/or triptans
* Patient had been using topiramate regularly

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2003-11; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Change in migraine days compared between the topiramate group and placebo group at the last 4 weeks of the open-label phase and the final 4 weeks of the placebo-controlled phase | Last 4 weeks of Open Label (OL) Phase and Double Blind (DB) Phase

SECONDARY OUTCOMES:
Patient's Satisfaction | Visit 6
  at the end of the OL Phase and at the end of the DB Phase
Health related quality of life as recorded in patient questionnaires (MIDAS and SF-12) | Visit 2, Visit 6, Visit 10
  At the start of the OL Phase; at the end of the of the OL Phase and at the end of the DB Phase
Health related quality of life as recorded in patient questionnaire (HIT-6) | Visit 2, Visit 4, Visit 6, Visit 8, Visit 10
  HIT-6 extra questioned at Week 8 and Week 34

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (68):
- Austria (2):
  - Innsbruck
  - Linz
- Belgium (4):
  - Antwerp
  - Charleroi
  - Leuven
  - Liÿge
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Czechia (2):
  - Hradec nad Svitavou
  - Prague
- Denmark (5):
  - Aabenraa
  - Esbjerg
  - Glostrup Municipality
  - Kÿbenhavn K
  - Odense
- France (6):
  - Colombes
  - Lille
  - Nice
  - Paris
  - Rouen
  - Voiron
- Germany (4):
  - Berlin
  - Essen
  - München
  - Mÿnster
- Greece (2):
  - Athens
  - Thessaloniki
- Hungary (4):
  - Budapest
  - Budapest Na
  - Miskolc
  - Szeged Na
- Ireland (2):
  - Cork
  - Dublin
- Norway (3):
  - Bodø
  - Oslo
  - Trondheim
- Poland (7):
  - Gdansk
  - Krakow Malopolska
  - Lodz
  - Mosina Poland
  - Poznan
  - Poznan Poland
  - Warsaw
- Portugal (3):
  - Coimbra
  - Lisbon
  - Porto
- Russia (2):
  - Moscow
  - Saint Petersburg
- Riyadh, Saudi Arabia
- Slovenia (2):
  - Ljubljana
  - Maribor
- Madrid, Spain
- Switzerland (3):
  - Biel/Bienne
  - Sankt Gallen
  - Zurich
- Turkey (Türkiye) (2):
  - Bursa
  - Istanbul
- United Kingdom (10):
  - Brighton
  - Glasgow
  - Helensburgh
  - Leicester
  - Newcastle upon Tyne
  - Northampton
  - Stoke-on-Trent
  - Sunderland
  - Surrey
  - York

REFERENCES:
- [Result] Diener HC, Agosti R, Allais G, Bergmans P, Bussone G, Davies B, Ertas M, Lanteri-Minet M, Reuter U, Sanchez Del Rio M, Schoenen J, Schwalen S, van Oene J; TOPMAT-MIG-303 Investigators Group. Cessation versus continuation of 6-month migraine preventive therapy with topiramate (PROMPT): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2007 Dec;6(12):1054-62. doi: 10.1016/S1474-4422(07)70272-7. Epub 2007 Nov 7. PMID 17988947
- See also: A double-blind, randomised, placebo-controlled, multicentre study to investigate the efficacy and tolerability of topiramate in prolonged migraine prevention. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=387&filename=CR003931_CSR.pdf